CLINICAL TRIAL: NCT06195865
Title: Autologous vs. Implant-based Breast Reconstruction: a Partially Randomised Patient Preference, Superiority Trial
Brief Title: Autologous vs. Implant-based Breast Reconstruction
Acronym: GoBreast II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-04754-01
Record Dates: First submitted 2023-12-21; First posted 2024-01-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Breast reconstruction; DIEP-flap; Implant-based breast reconstruction
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Randomised DIEP flap (Active Comparator)
  Interventions: Procedure: DIEP-flap
- Randomised implant-based (Active Comparator)
  Interventions: Procedure: Implant
- Preference DIEP-flap (Active Comparator)
  Interventions: Procedure: DIEP-flap
- Preference implant-based (Active Comparator)
  Interventions: Procedure: Implant

INTERVENTIONS:
Procedure: DIEP-flap — Breast reconstruction with a deep inferior epigastric perforator flap
  Arms: Preference DIEP-flap; Randomised DIEP flap
Procedure: Implant — Breast reconstruction with an implant-based technique
  Arms: Preference implant-based; Randomised implant-based

SUMMARY:
Although breast reconstruction is an integral part of breast cancer treatment, there is little high-quality evidence to indicate which method is the most effective. The objective of this study is to compare implant-based and autologous breast reconstruction, in non-radiated patients. The primary outcome is patient reported breast-specific quality of life/satisfaction and the secondary outcomes are complications, factors affecting satisfaction, and cost-effectiveness. Moreover, the study aims to improve the evidence for trial decision-making in breast reconstruction. Randomized controlled trials (RCT) are generally thought to provide the most solid scientific evidence, but there are significant barriers to conducting RCTs in breast reconstruction, making both recruitment and achieving unbiased and generalisable results a challenge. The study design partially randomised patient preference trial (RPPT) might be a way to overcome these challenges. In the present study, patients who consent to randomisation will be randomised to implant-based and autologous breast reconstruction, whereas patients with strong preferences will be able to choose method. The study is designed as a superiority trial based on BREAST-Q and 124 participants will be randomised. In the preference cohort patients will be included until 62 participants have selected the least popular alternative. Follow-up will be 60-months. Embedded qualitative studies and within-trial economic evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Biological female
* >18 years of age
* American Society of anesthesiologist classification (ASA) 1-2
* Patient must have had or be scheduled for a mastectomy
* Ability to give informed consent
* Ability to communicate in Swedish

Exclusion Criteria:

* ASA > 2
* BMI > 30 kg/m2
* Smoking1 radiotherapy to the breast in question.
* Radiotherapy is expected post-operatively.
* Locally advanced breast cancer
* Metastasised breast cancer
* Comorbidity and/or drugs that affect wound healing.
* Unstable psychiatric co-morbidity
* Abdominal scaring/chest scaring making a DIEP/implant-based reconstruction unsuitable

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological females.
Enrollment: 250 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with the breast/s and breast-specific quality of life | 5 years
  Satisfaction with the breast/s and breast-specific quality of life measured with BREAST-Q reconstruction.The patient rates all items on 3-, 4-, and 5-point Likert-scales. A raw score, that is converted to a score 0-100, is calculated for each domain. A higher score indicates a greater satisfaction or better quality of life.
Cost-effectiveness | 5 years+ simulation model based on 20 years
  The net cost divided for society by changes in health outcomes measured with Breast-Q and EQ5D.

SECONDARY OUTCOMES:
Complications | 5 years
  Complications classified as types and according to the Clavien-Dindo Classification (CDC) of surgical complications. According to CDC all complications are graded from 1 (any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions) to 5 (Patient demise). Comprehensive Complication Index (CCI) scores will also be used. The CCI is calculated from CDC as the sum of all complications that are weighted for their severity, yielding a scale from 0-100. A higher CCI means more severe and more complications. All participating surgeons will be given a list of study specific definitions of complications.
Surgical revisions | 5 years
  All operations performed will be recorded and classified according to the international classification of disease in the operation planing program Orbit.
Satisfaction with the donor-site | 5 years
  Satisfaction with the donor site will be measured with the abdominal domain of Breast-Q.The patient rates all items on 3-, 4-, and 5-point Likert-scales. A raw score, that is converted to a score 0-100, is calculated for each domain. A higher score indicates a greater satisfaction or better quality of life.
Symptoms of depression and anxiety | 5 years
  Symptoms of depression and anxiety will be measured with the Hospital Anxiety and Depression Scale (HADS).The HADS is a fourteen item scale that generates: Seven of the items relate to anxiety and seven relate to depression.For both scales, scores of less than 7 indicate non-cases. 8-10 mild, 11-14 moderate, 15-21 severe.
Body image | 5 years
  Body image will be measured with the Multidimensional Body-Self Relation Questionnaire (MBSRQ).Multidimensional body-self relations questionnaire- appearance scales.It is a 34-item self-report questionnaire designed to measure appearance related components of body-image. In consists of five subscales: appearance evaluation, appearance orientation, body areas satisfaction, overweight preoccupation, and self-classified weight. It is a 5-point Likert-scale ranging from 1 to 5.
Body investment | 5 years
  Body investment will be measured with the Appearance Schemas Inventory-revised (ASI-R).Appearance schemas inventory-revised: is a 20-item self-report questionnaire designed to measure body-image investment. It consists of two subscales, self-evaluative salience (SES) and motivational salience (MS). It is a 5-point Likert-scale ranging from 1 (strongly disagree) to 5 (strongly agree). Twelve items relate to SES and eight items relate to MS. The total score is the mean of the 20 items, and the score of the subscales is the mean of the items relating to each subscale. A high score indicates greater body-image investment.
Generic quality of life | 5 years
  Generic quality of life will be measured with EuroQoL-5 dimensions (EQ-5D-3L).n EQ-5D-3L, the five dimensions each have three response levels of severity.Respondents are asked to choose the statement in each dimension that best describes their health status on the day they are surveyed. Their responses are coded as a number (1, 2, or 3) that corresponds to the respective level of severity: 1 indicates no problems, 2 some problems, and 3 extreme problems.

OTHER OUTCOMES:
Expectations | Pre-op
  Pre-operative expectations will be measured with the BREAST-Q expectations domain. The patient rates all items on 3-, 4-, and 5-point Likert-scales. A raw score, that is converted to a score 0-100, is calculated for each domain. A higher score indicates a greater satisfaction or better quality of life.
Patient's goals with the reconstruction | Pre-op
  patient's goals with the reconstruction will be documented using the PEGASUS instrument. Patients' Expectations and Goals of reconstruction. Assisting Shared Understanding of Surgery) tool to make the decision of whether they want a breast reconstruction. The tool is used to form a basis for a patient-centred dialogue around breast reconstruction.
Study with a trial (SWAT):The choice of breast reconstruction and the choice of reconstructive method. | Longitudinal - the same participants will be interviewed at allocation and 12 months after the reconstruction.
  Qualitative study - participants will be recruited from the preference cohort.
Study with a trial (SWAT):What makes a participant very satisfied or very dissatisfied. | 12 months after reconstruction
  Qualitative study -Participants will be recruited from both cohorts among women who scored high/low, compared to the mean, on BREAST-Q outcome and satisfaction with breast/s.
Study with a trial (SWAT): Experiences with the trial process. | Different participants from both cohorts are interviewed at allocation, 3 and 12 months to explore if there are different themes at different time points.
  Qualitative study -How the participant experienced the trial process, how it can be ameliorated to increase recruitment, retention, and follow-up rates of questionnaires and how participation information leaflet should be designed/written to maximize recruitment.
Differences between the preference and the randomized cohort | Preoperatively and 12 months after reconstruction
  Differences regarding demographic factors as well as pre-operative satisfaction with breasts, expectations, body-image, symptoms of depression and anxiety, and generic quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska university hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansson E, Lofstrand J, Larsson C, Uusimaki A, Svensson K, Ekman A, Svensson M, Paganini A. Gothenburg Breast reconstruction (GoBreast) II protocol: a Swedish partially randomised patient preference, superiority trial comparing autologous and implant-based breast reconstruction. BMJ Open. 2024 Jul 17;14(7):e084025. doi: 10.1136/bmjopen-2024-084025. PMID 39019639